CLINICAL TRIAL: NCT00830141
Title: Study of the Molecular Basis in the Pathophysiology of Food Intake and Growth in Children
Acronym: Ghrelin
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Yardena Tenenbaum-Rakover, Head of Pediatric Endocrinology, HaEmek Medical Center, Israel
Other Study IDs: 0040-08-EMC
Record Dates: First submitted 2009-01-25; First posted 2009-01-27 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Obesity; Short Stature
Keywords: Ghrelin; obesity; idiopathic short stature (ISS)
MeSH Terms: conditions — Obesity; Dwarfism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA will be isolated from peripheral blood by standard methods. The corresponding intron-exon boundaries of ghrelin and GHSR genes will be analyzed by direct sequencing using the ABI Prism 3100 DNA Analyzer
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: 50 children with GH deficiency
- 2: 50 children with ISS
- 3: 50 children with FTT
- 4: 50 children with obesity
- 5: 50 children without short stature or obesity will serve as controls

SUMMARY:
Obesity, now a global epidemic, is a leading cause of illness and mortality in the developed world. To better understand the pathophysiological mechanisms that underlie weight disorders, increasing attention is being paid to central regulatory elements in energy homeostasis, including food intake and energy expenditure. The human hormone ghrelin is secreted as a preprohormone (preproghrelin), from which two hormones with antagonistic effects are derived: ghrelin, which has orexigenic effects and obestatin, which has anorexigenic effects. Ghrelin's actions are mediated by GH secretagogue receptor (GHSR). Ghrelin synthesis occurs predominantly in epithelial cells of the fundus of the stomach. . As the ligand for GHSR, ghrelin stimulates secretion of GH. In both rodents and humans, ghrelin regulates hunger though its action on hypothalamic feeding centers. Other effects of ghrelin include stimulating gastric emptying, positive effects on cardiovascular function, increasing intestinal peristalsis, and positive exocrine and paracrine pancreatic secretion. Despite its important physiological role, its precise regulatory mechanisms remain ambiguous. Thus, it has been suggested that mutations in ghrelin and its receptor will present clinically with obesity, eating disorders or growth disturbances. To date, only four different mutations have been reported in GHSR and no mutations have been found in the ghrelin gene.

Working hypothesis and aims: We hypothesize that mutations in ghrelin or in its receptor, GHSR, affect appetite regulation and cause growth and eating disorders.

DETAILED DESCRIPTION:
Background: Obesity, now a global epidemic, is a leading cause of illness and mortality in the developed world. To better understand the pathophysiological mechanisms that underlie weight disorders, increasing attention is being paid to central regulatory elements in energy homeostasis, including food intake and energy expenditure. The human hormone ghrelin is secreted as a preprohormone (preproghrelin), from which two hormones with antagonistic effects are derived: ghrelin, which has orexigenic effects and obestatin, which has anorexigenic effects. Ghrelin's actions are mediated by GH secretagogue receptor (GHSR). Ghrelin synthesis occurs predominantly in epithelial cells of the fundus of the stomach. . As the ligand for GHSR, ghrelin stimulates secretion of GH. In both rodents and humans, ghrelin regulates hunger though its action on hypothalamic feeding centers. Other effects of ghrelin include stimulating gastric emptying, positive effects on cardiovascular function, increasing intestinal peristalsis, and positive exocrine and paracrine pancreatic secretion. Despite its important physiological role, its precise regulatory mechanisms remain ambiguous. Thus, it has been suggested that mutations in ghrelin and its receptor will present clinically with obesity, eating disorders or growth disturbances. To date, only four different mutations have been reported in GHSR and no mutations have been found in the ghrelin gene.

Working hypothesis and aims: We hypothesize that mutations in ghrelin or in its receptor, GHSR, affect appetite regulation and cause growth and eating disorders.

Methods: A total of 250 children followed in the pediatric endocrine department at Ha'Emek Medical Center will be divided into four groups: 50 children with GH deficiency, 50 obese children, 50 children with failure to thrive (FTT),and 50 children with idiopathic short stature (ISS). In addition, 50 children without growth or weight disorders will be included as a control group.

Genomic DNA will be isolated from the peripheral blood by standard methods. The corresponding intron-exon boundaries of the ghrelin and GHSR genes will be analyzed by direct sequencing using an ABI Prism 3100 DNA Analyzer.

Expected results: We anticipate that mutations in ghrelin or its receptor will affect growth and appetite regulation.

Importance: The findings of this study will expand our understanding of ghrelin's role in growth and appetite regulation.

Probable implications for medicine: The development of more specific therapeutic modalities for the treatment of short stature and obesity in children may become possible.

ELIGIBILITY:
Inclusion Criteria:

* Group1: Children with GH deficiency diagnosed by 2 provocative tests with peak GH less than 10 ng/ml.
* Group 2:Children with height less than the 3rd centile without any etiology
* Group 3:children with failure to thrive until the age of 3 years.
* Group 4: children with obesity defined by BMI above the 90th centile for age and sex.
* Group 5: children with no endocrine diseases and without obesity or short stature.

Exclusion Criteria:

* Children with known pediatric or endocrine diseases.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 250 children followed in the pediatric endocrine department at Ha'Emek Medical Center will be divided into 5 groups: 50 children with GH deficiency,50 obese children, 50 children with failure to thrive (FTT)and 50 children with idiopathic short stature (ISS). 50 children without growth and weight disorders will be included as a control group.
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yardena Tenenbaum-Rakover, MD, Principal Investigator — Ha"Emek Medical Center, Afula, ISRAEL